CLINICAL TRIAL: NCT05290064
Title: Effect of Ultra-processed Versus Unprocessed Diets on Energy Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 220002; 22-DK-0002
Record Dates: First submitted 2022-03-19; First posted 2022-03-22 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08-21

CONDITIONS: Healthy Diet; Obesity
Keywords: Body Weight; Food Intake; Fat; Calories; Body Mass Index
MeSH Terms: conditions — Obesity; Body Weight; Platelet Glycoprotein IV Deficiency | interventions — Food, Processed

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1/UPF HH, UPF HL, UNF LL, UPF LL (Experimental): Four diets in the order specified
  Interventions: Other: Ultra-processed food, high energy density; Other: Ultra-processed food, both low; Other: Ultra-processed food, both high; Other: Unprocessed food diet
- 2/ UPF HL, UPF LL, UPF HH, UNF LL (Experimental): Four diets in the order specified
  Interventions: Other: Ultra-processed food, high energy density; Other: Ultra-processed food, both low; Other: Ultra-processed food, both high; Other: Unprocessed food diet
- 3/ UPF LL, UNF LL, UPF HL, UPF HH (Experimental): Four diets in the order specified
  Interventions: Other: Ultra-processed food, high energy density; Other: Ultra-processed food, both low; Other: Ultra-processed food, both high; Other: Unprocessed food diet
- 4/ UNF LL, UPF HH, UPF LL, UPF HL (Experimental): Four diets in the order specified
  Interventions: Other: Ultra-processed food, high energy density; Other: Ultra-processed food, both low; Other: Ultra-processed food, both high; Other: Unprocessed food diet

INTERVENTIONS:
Other: Ultra-processed food, high energy density — Ultra-processed diet that is high in non-beverage energy density and low in hyperpalatable foods
Other: Ultra-processed food, both low — Ultra-processed diet that is low in both non-beverage energy density and hyperpalatable foods
Other: Ultra-processed food, both high — Ultra-processed diet that is high in both non-beverage energy density and hyperpalatable foods
Other: Unprocessed food diet — Unprocessed diet that is low in both non-beverage energy density and hyperpalatable foods

SUMMARY:
Protocol Number: 22DK0002

Title: Effects of Ultra-processed versus Unprocessed Diets on Energy Metabolism

Background:

Many diets worldwide include both processed and unprocessed foods. Researchers want to study the effects these foods have on a person s health.

Objective:

To study how different diets affect a person s health and metabolism.

Eligibility:

Adults aged 18 60 without diabetes who have stable weight and can exercise.

Design:

Participants will be screened with:

Medical history

Physical exam

Heart tests

Resting energy expenditure (to determine calorie needs)

Blood and urine tests

20-minute stationary bicycle session

Food, diet, and mental health questionnaires

Participants will stay at NIH for 4 weeks. They will receive 3 meals a day and may eat as little or as much as they want. The diet will change each week. Their weight will be recorded daily. They will ride a stationary bicycle daily. Each week, they will do the following:

Spend 1 day in a special room that assesses their metabolism

Have 24-hour urine collections

Give skin and fecal samples

Repeat some screening tests

Have scans to measure body fat

Complete computerized behavior tasks

Wear an activity monitor to track physical activity

Wear a glucose monitor. A sensor will be inserted under the skin with a small needle. It will be replaced weekly.

Take taste tests. They will swish water and flavored liquids around in their mouth and pick which ones had a non-neutral taste. They will also compare liquids for which ones taste better.

Participation will last for 4 weeks.

Sponsoring Institution: National Institute of Diabetes and Digestive and Kidney Diseases

...

DETAILED DESCRIPTION:
This is a randomized crossover study of adult volunteers to determine the health effects of four different diets varying in non-beverage energy density, hyperpalatable foods, as well as the degree, extent, and purpose of processing according to the NOVA classification system.

Objectives/Endpoints:

Primary Aim:

To determine differences in health effects during four 1-week test diets.

Secondary Aims:

To determine differences in mean eating rate (grams per minute) and palatability of meals between the four 1-week test diets.

Exploratory Aims:

Several exploratory measurements are planned to help comprehensively phenotype the effects of the test diets and are intended to be hypothesis-generating.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Provision of signed and dated informed consent form
* Adults age 18-60 years, male and female
* Weight stable (< +/- 5 % body weight change over past 6 months) as determined by volunteer report
* Body mass index (BMI) > =20 kg/m2
* Body weight > = 53 kg
* Able to complete daily bouts of stationary cycling at a moderate rate and intensity with a HR equal to or greater than 0.3(SqrRoot) (220-age-HRrest)+HRrest but not exceeding 0.4(SqrRoot) (220-age-HRrest)+HRrest and no signs of arrhythmia
* Willingness to comply with all study procedures and Lifestyle Considerations for the duration of the study per the discretion of the PI.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Evidence of diseases or conditions that may influence appetite (e.g., cancer, diabetes, alterations of smell or taste post COVID-19), or other conditions at the discretion of the PI and/or study team).
* Taking prescription medications or other drugs that may influence appetite (including, but not limited to, diet/weight-loss medication or other medications at the discretion of the PI and/or study team)
* Positive pregnancy test or lactation as determined by volunteer report (women only)
* Participating in a regular exercise program (> 2h/week of vigorous activity) as determined by volunteer report
* Hematocrit < 37% (women only)
* Hematocrit < 40% (men only)
* Caffeine consumption > 300 mg/day as determined by volunteer report
* Alcohol consumption > 3 drinks per day for men or > 2 drinks per day for women as determined by volunteer report
* Regular use of tobacco (smoking or chewing), amphetamines, cocaine, heroin, or marijuana over past 6 months as determined by volunteer report. Subjects may also be excluded based on a urine drug test.
* Psychological conditions as determined by volunteer report such as (but not limited to) eating disorders, depression, bipolar disorders, that would be incompatible with safe and successful participation in this study, as determined by investigators
* Volunteers with strict dietary concerns (e.g. vegetarian or kosher diet, food allergies) or a reported dislike of a significant fraction of the study foods
* Volunteers unwilling or unable to give informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2022-11-04 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Energy Metabolism (kcal per day) | Four 1-week diets
  Energy Metabolism averaged over 7 days for each diet, measured in kilocalories (kcal) per day. Primary comparisons will be between UPF HH & UPF HL, UPF HL & UPF LL, UPF LL & UNF LL, UPF HH & UNF LL.

SECONDARY OUTCOMES:
Meal eating rate (grams per minute) | Four 1-week diets
  This will be determined by the measured duration of the meals along with the measured mass of food consumed.
Meal palatability | Four 1-week diets
  This will be measured via questionnaires using visual analogue scales.

CONTACTS AND LOCATIONS:
Overall Officials: Valerie L Darcey, Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2022-DK-0002.html